CLINICAL TRIAL: NCT06322277
Title: The Regional Pediatric Network and the Use of Low-cost Molecular Diagnostic Techniques Cost as a New Management and Surveillance Model for Diseases Preventable by Vaccinations.
Brief Title: Use of Low-cost Molecular Diagnostic Techniques as a New Surveillance Model for Diseases Preventable by Vaccinations.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Massimo Resti, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NETVAC
Record Dates: First submitted 2024-02-28; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with viral/bacterial infection (Other)
  Interventions: Other: Analysis of biological sample

INTERVENTIONS:
Other: Analysis of biological sample — Confermation of type of infection with RT-PCR.

SUMMARY:
Vaccine-preventable disease (VPD) surveillance should be a priority throughout the world. In Italy, however, there is limited attention to the epidemiology of VPDs, with the consequence that their incidence is largely underestimated. Although notification of vaccine-preventable diseases is mandatory, very often the etiologic agents causing VPDs are not identified the etiological agents causing the major and most severe infectious diseases in childhood. Several reasons underlie the underestimation. For example, not having a good surveillance system does not allow us to organize a sustainable prevention project for example based on on the introduction of new vaccinations. For example the limited use of low-cost high-sensitivity techniques such as real-time PCR, which could, if more widely used, improve pathogen identification with 3 times the sensitivity of standard cultural methods. Therefore, the idea of this multicenter, biological sample study is to take advantage of the regional pediatric network with the goal of improving VPD surveillance and increase awareness of the importance of surveillance of preventable diseases with the vaccine within the pediatric network.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 0-18 years with infectious disease (bacterial or viral) diagnosed by molecular techniques at the AOU Meyer Immunology Laboratory
* Obtaining informed consent

Exclusion Criteria:

* Individuals with concomitant diseases such as cystic fibrosis, known immunodeficiency, or with infection suspected nosocomial (hospitalization or hospital admission within 15 days prior to the onset of symptoms) will be excluded from the study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of major VPDs (vaccine-preventable infectious diseases): pertussis, influenza virus, respiratory syncytial virus, S.pneumoniae, N.meningitidis, H.influenzae. | After 3 years from the beginning of the study
  Molecular surveillance data analysis of pertussis, respiratory virus disease, invasive bacterial diseases. We will measure the incidence rate of predictable disease with vaccination, stratifying by biological sex, age, other risk factors, and severity of infection during the project.
  (IBD) due to capsule bacteria (Streptococcus pneumoniae, Neisseria meningitidis, Haemophilus influenzae) and other vaccine-preventable infections (e.g., viral flu)

SECONDARY OUTCOMES:
Frequency of principal serotype, serogroups of pathogens causative for VPDs. | After 3 years from the beginning of the study
  Analysis of molecular characteristics of germs identified in pediatric subjects with VPDs.
Number of meeting to diffuse the NETVAC results in Tuscany network. | After 3 years and 6 months from the beginning of the study
  Expand and spread knowledge of the importance of active and molecular surveillance in the pediatric network consisting of hospital centers and family pediatricians in Tuscany through the organization of at least two meetings/year for three years between centers hospitals in Tuscany, family pediatricians within the regional pediatric network and pediatric scientific societies in order to disseminate the role of molecular diagnosis in the active surveillance against vaccine-preventable infectious diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Resti, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (4):
- Italy (4):
  - Ospedale San Donato, Arezzo
  - Immunology Laboratory Meyer Children's Hospital, IRCCS, Florence
  - Meyer Children's Hospital IRCCS, Florence
  - UO Pediatria Universitaria Ospedale S.Chiara, Pisa